CLINICAL TRIAL: NCT03776318
Title: A Multicenter, Randomized, Follow-up Study to Evaluate the Long-Term Safety of Clonidine Micropellets for the Treatment of Pain Associated With Lumbosacral Radiculopathy in Adults
Brief Title: Long-Term Follow-up Safety of Clonidine Micropellets
Acronym: RePRIEVE-CM-LT
Status: Completed | Type: Observational
Sponsor: Sollis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STX-015-18-02
Record Dates: First submitted 2018-12-01; First posted 2018-12-14 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Lumbosacral Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Safety Group: STX-015-18-01 Clonidine Micropellet long-term safety follow-up
  Interventions: Drug: Long-Term Safety Follow-up
- Sham Control: STX-015-18-01 Sham control long-term safety follow-up
  Interventions: Drug: Long-Term Safety Follow-up

INTERVENTIONS:
Drug: Long-Term Safety Follow-up — STX-015-18-01 long-term safety follow-up

SUMMARY:
Long-term follow-up study to evaluate the safety of clonidine micropellets up to 12 months post injection.

ELIGIBILITY:
Inclusion Criteria:

* Subject who have successfully completed all STX-015-18-01 study related activities, are reconfirmed to be eligible and have signed informed consent to participate.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, have demonstrated significant non-compliance with STX-015-18-01 study procedures.
* Subjects who were unblinded to their treatment in STX-015-18-01 study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comprised of the first 100 subjects who completed all STX-015-18-01 study-related activities, age 18-70, male/female, reconfirmed eligible and signed informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Average and Worst NRS from Day 60 post injection to 12 months post injection | 10 months from completing Day 60 of the STX-015-18-01 study
  Difference in NRS pain scores from Day 60 of STX-015-18-01 to month 12 post injection

SECONDARY OUTCOMES:
Incidence of Surgeries | 12 months from day of injection
  Difference in incidence of surgery, invasive treatment, and prescription medications due to radicular leg pain from Day 30 post injection to month 12 post injection from a cohort of subjects completing STX-015-18-01.
Incidence of Invasive treatment received | 12 months from day of injection
  Difference in incidence of invasive treatment due to radicular leg pain from Day 30 post injection to month 12 post injection from a cohort of subjects completing STX-015-18-01
Number of Prescription medications taken | 12 months from day of injection
  Difference in incidence of invasive treatment due to radicular leg pain from Day 30 post injection to month 12 post injection from a cohort of subjects completing STX-015-18-01

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gilligan, MD, Principal Investigator — Brigham and Women's Hospital
Locations (25):
- United States (25):
  - Sollis Clinical Study Site 36, Mobile, Alabama
  - Sollis Clinical Study Site 44, Phoenix, Arizona
  - Sollis Clinical Study Site 40, Tucson, Arizona
  - Sollis Clinical Study Site 49, Rancho Mirage, California
  - Sollis Clinical Study Site 30, Washington D.C., District of Columbia
  - Sollis Clinical Study Site 35, Fort Lauderdale, Florida
  - Sollis Clinical Study Site 38, Miami, Florida
  - Sollis Clinical Study Site 12, Bloomington, Illinois
  - Sollis Clinical Study Site 13, Chicago, Illinois
  - Sollis Clinical Study Site 14, Kansas City, Kansas
  - Sollis Clinical Study Site 37, Overland Park, Kansas
  - Sollis Clinical Study Site 10, Edgewood, Kentucky
  - Sollis Clinical Study Site 15, Brookline, Massachusetts
  - Sollis Clinical Study Site 17, Shrewsbury, New Jersey
  - Sollis Clinical Study Site 31, Rochester, New York
  - Sollis Clinical Study Site 18, Winston-Salem, North Carolina
  - Sollis Clinical Study Site 21, Cleveland, Ohio
  - Sollis Clinical Study Site 33, Cleveland, Ohio
  - Sollis Clinical Study Site 19, Edmond, Oklahoma
  - Sollis Clinical Study Site 46, Eugene, Oregon
  - Sollis Clinical Study Site 42, Dallas, Texas
  - Sollis Clinical Study Site 34, Houston, Texas
  - Sollis Clinical Study Site 47, Salt Lake City, Utah
  - Sollis Clinical Study Site 23, Morgantown, West Virginia
  - Sollis Clinical Study Site 27, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No